CLINICAL TRIAL: NCT03956485
Title: Multicentre Registry of Patients With Spontaneous Acute Intracerebral Hemorrhage in Catalonia
Brief Title: Multicentre Registry of Patients With Spontaneous Acute Intracerebral Hemorrhage in Catalonia (HIC-CAT).
Acronym: HIC-CAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fundació Ictus (Unknown); Pla Director de la Malaltia vascular Cerebral, Departament de Salut (Unknown)
Responsible Party: Sponsor
Other Study IDs: IIBSP-HIC-2019-22
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Intracerebral Hemorrhage
Keywords: intracerebral hemorrhage; outcome; transportation; transfer; prognosis
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Type of center — Tertiary versus non-tertiary
  Other Names: Time from onset to admission

SUMMARY:
A population-based registry in Catalonia of patients with acute spontaneous Intracerebral Hemorrhage, to investigate whether type of center and time from onset to admission is associated with functional outcome and mortality.

DETAILED DESCRIPTION:
Introduction. Recent studies show that there are potentially beneficial therapeutic measures for the patient with acute intracerebral hemorrhage (ICH), which should be applied urgently and that some would only be available in tertiary stroke centers (TSC). However, the transportation criteria for ICH patients are not well defined.

Objectives: Design and implementation of a registry (HIC-CAT) of patients with HIC in the healthcare network of public hospitals in Catalonia, which does not modify the current logistics but collects data related to patients and TSC, interhospital transfers and non-TSC centers. The registry will allow us to evaluate the hypothesis that: 1) Patient care in TSC decreases the probability of death or dependence in patients with spontaneous ICH compared to non-TSC; and 2) The shorter the time until admission to a TSC, the better the survival and functional outcome. This will be due to the application of diagnostic, therapeutic and structural measures at the TSC. In addition, organ donation will be more frequent in a TSC.

Methods: Observational, prospective, multicentre, population study of 2500 consecutive patients with spontaneous ICH of less than 24 hours from the onset of symptoms and Rankin scale score 0-3. We will collect times, clinical and radiological variables, vital and functional outcome at 3 months follow-up. Number of organ donations. Primary variable: Functional outcome at 3 months (Rankin 0-3). Statistics: Multivariate analysis with logistic regression, propensity matching scores.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of spontaneous intracerebral hemorrhage who is diagnosed in any of the participant hospitals

Exclusion Criteria:

* Traumatic intracerebral hemorrhage
* >24 hours from onset to admission
* Prior Rankin scale score >3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of acute spontaneous intracerebral hemorrhage in Catalonia during a period of 2 years
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 3 months after onset
  Rankin scale score, favourable if 0,1, 2 or 3

SECONDARY OUTCOMES:
Mortality | 3 months
  mortality within the first 3 months after onset
Hematoma expansion | 72 hours
  increase in hematoma volume (>33% and/or 6 ml) from baseline CT to follow-up CT
Stroke Unit admission | 3 months
  Percentage of patients admitted to a stroke unit
Neurological worsening | During admission
  increase in 4 or more points in the NIHSS score and/or decrease >1 point in the Glasgow coma scale score

CONTACTS AND LOCATIONS:
Locations (26):
- Spain (26):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Fundació Hospital Asil Granollers, Granollers, Barcelona
  - Hospital d'Igualada, Igualada, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Moisés Broggi, Sant Joan Despí, Barcelona
  - Mutua de Terrassa, Terrassa, Barcelona
  - Hospital de Figueras, Figueras, Girona
  - Hospital de Palamós, Palamós, Girona
  - Fundació Sant hospital de la Seu d'Urgell, La Seu d'Urgell, Lleida
  - Hospital de Tremp, Tremp, Lleida
  - Hospital de la Cinta, Tortosa, Tarragona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Consorci Sanitari del Garraf, Barcelona
  - Hospital Clínic, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Dr Josep Trueta, Girona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital de la Cerdanya, Lleida
  - Centre Hospitalari Althaia, Manresa
  - Hospital Comarcal Móra d'Ebre, Móra d'Ebre
  - Hospital joan XXIII, Tarragona
  - Hospital de Vic, Vic
  - Hospital de Vilafranca, Vilafranca del Penedès

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lambea-Gil A, Marti-Fabregas J, Cardona P, Rodriguez-Luna D, Millan M, Amaro S, Prats-Sanchez L, Silva Y, Sero L, Rodriguez-Campello A, Canovas D, Martinez-Domeno A, Guasch-Jimenez M, Ezcurra-Diaz G, Carcel-Marquez J, Fernandez-Cadenas I, Perez De La Ossa N, Abilleira S, Salvat-Plana M, Fagundez O, Camps-Renom P, Ramos-Pachon A; as the HIC-CAT investigators. Effect of Onset-to-Admission Time and Care Bundle Achievement on Functional Outcomes in Patients With ICH: A Population-Based Study. Neurology. 2025 Oct 21;105(8):e214176. doi: 10.1212/WNL.0000000000214176. Epub 2025 Sep 30. PMID 41026995
- [Derived] Marti-Fabregas J, Ramos-Pachon A, Prats-Sanchez L, Nunez-Guillen A, Rodriguez BL, Rodriguez-Luna D, Amaro S, Silva Y, Rodriguez-Campello A, Puig I, Gomez-Choco M, Vazquez-Justes D, Guanyabens N, Cocho D, Canovas D, Steinhauer EG, Llull L, Guasch-Jimenez M, Martinez-Domeno A, Marin R, Lambea-Gil A, Diaz GE, Paipa-Merchan A, Quesada H, Casadevall MP, Wenger D, Pancorbo O, Sero L, Perez J, Costa X, Zaragoza J, Rodriguez-Villatoro N, Catena E, Calvo NM, Krupinski J, De La Ossa NP, Abilleira S, Salvat-Planas M, Fagundez O, Camps-Renom P; for HIC-CAT. Influence of Hospital Type on Outcomes of Patients With Acute Spontaneous Intracerebral Hemorrhage: A Population-Based Study. Neurology. 2024 Jul 23;103(2):e209539. doi: 10.1212/WNL.0000000000209539. Epub 2024 Jun 14. PMID 38875516